CLINICAL TRIAL: NCT03485560
Title: Revitalization of Damaged Sking Due to Chronic Skin Diseases
Brief Title: Revitalization of Damaged Skin Due to Chronic Skin Diseases
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ace Cells Lab Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACEcsd
Record Dates: First submitted 2017-10-07; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2017-11

CONDITIONS: Chronic Eczema; Psoriasis; Atopic Dermatitis
Keywords: chronic skin disease; psoriasis; Eczema; atopic dermatitis
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- internvention of Chrinic skin conditions (Experimental): All cases of chronic skin conditions will be included to measure the effect on the 3 of them and whihc one will respond to the treatment better
  Interventions: Combination Product: ACE CSD

INTERVENTIONS:
Combination Product: ACE CSD — Topical application of the ACE CSD 4 times daily.
  Other Names: ACE Skin immune

SUMMARY:
Chronic skin disease lead to skin damage and disfiguring to the patient skin. Sometimes, achieving normal skin is not possible by the normal traditional treatment, this study is focusing on use of ACE CSD formula which is mixture of natural peptides and herbs. the main aim is to restore the normal skin appearance for the patient and control the episodes of flare.

DETAILED DESCRIPTION:
Psoriasis is a chronic, immune mediated (type 2 and type 17) chronic skin disease. The production of the immune proteins that leads to continuous inflammatory mediated process. The result of chronic inflammation is they hyper keratotic layer of skin which gets attacks of atopic dermatitis leading to symptoms of itching, pruritis and in situ bleeding.

ACE CSD, with the multiple factors that mediates the immune response and control the protein receptors, in addition to the multiple regeneration peptides that are specifically extracted from healthy skin of newly born sheep; in addition to multiple Chinese herbs that contains different anabolic factors was tested to be able to regenerate the damaged skin and locally modulate the immunity reactions so the skin can regenerate fully to replace the damaged skin with normal healthy skin.

ELIGIBILITY:
Inclusion Criteria:

* Chronic skin condition lasts for more than 1 year.
* tried traditional treatment with limited or without effect.
* not on steroids for at least 6 weeks.

Exclusion Criteria:

* patients on steroid.
* patients intolerable to protein or allergic to proteins
* during pregnancy or lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Regeneration of the damaged skin lesion | 6 - 9 months
  Complete regeneration of the affected skin lesions from the skin disease.

SECONDARY OUTCOMES:
Flare control | 1-3 months
  During the attacks of flare, the regenerated skin does not get affected nor show erythematous reaction

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Diana Diana, MSc Dermatology, Principal Investigator — ACE cells Lab europe DOO
Locations (2):
- ACE cells Lab Europe Doo, Belgrade, Serbia
- ACE Cells Lab Limited, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No